CLINICAL TRIAL: NCT01855087
Title: A Study of Safety and Efficacy of Sitagliptin Added to Insulin Therapy in the Treatment of Type 2 Diabetes in Kanagawa
Brief Title: Safety and Efficacy of Sitagliptin Added to Insulin Therapy for Type 2 Diabetes
Acronym: ASSIST-K
Status: Completed | Type: Observational
Sponsor: Kanagawa Physicians Association (Other)
Collaborators: The Japan Kidney Foundation (Other)
Responsible Party: Principal Investigator, Ikuro Matsuba, Chairperson, Kanagawa Physicians Association
Other Study IDs: R875
Record Dates: First submitted 2013-05-10; First posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
There is paucity of information about the combination therapy with dipeptidyl peptidase-4 inhibitor sitagliptin and insulin. This study aimed to retrospectively investigate the safety and efficacy of this therapeutic modality in Japanese patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* outpatients with type 2 diabetes
* addition of sitagliptin to insulin therapy
* aged 20 years or older
* HbA1c of 6.9% or higher (NGSP) at the time of adding sitagliptin

Exclusion Criteria:

* history of hypersensitivity to sitagliptin
* severe ketosis, diabetic coma, and/or precoma within 6 months before sitagliptin administration
* sever infection and/or severe trauma, and/or patients who are scheduled to undergo / have recently underwent surgery
* severe renal dysfunction (serum creatinine [mg/dL]: 2.5 or higher for men; 2.0 or higher for women)
* ongoing treatment with glinide(s)
* judgment as ineligible for the study by the attending physician

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: One-thousand Japanese patients with type 2 diabetes
Sampling Method: Non-Probability Sample
Dates: Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Blood glucose level | Six months after starting sitagliptin-insulin combination therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Takai Naika Clinic, Kamakura, Kanagawa, Japan